CLINICAL TRIAL: NCT05812313
Title: Educators and Young People's Mental Health During Their Vocational Education in the Health and Care Professions - a Cross-Sequential Observational Study
Brief Title: Educators and Young People's Mental Health
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Manuel Stadtmann (Other)
Collaborators: Berufs- und Weiterbildungszentrum für Gesundheits- und Sozialberufe St.Gallen (BZGS) (Unknown)
Responsible Party: Sponsor-Investigator, Manuel Stadtmann, Prof. Dr. Manuel P. Stadtmann, St.Gallen University of Applied Sciences
Organization: St.Gallen University of Applied Sciences (Other)
Other Study IDs: youcoment_0001
Record Dates: First submitted 2023-02-16; First posted 2023-04-13 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Mental Health Issue; Adolescent Development; Mental Health Wellness 1; Mental Health Wellness 2; Mental Disorder in Adolescence; Social Stigma
Keywords: adolescent; health promotion; mental health; schools; health literacy; cross sectional; educators; vocational education; health care profession; social care professions
MeSH Terms: conditions — Social Stigma; Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- vocational trainees in health and care professions
- vocational educators in health and care professions.

SUMMARY:
The aim of the present study is to assess the current state of mental health of educators and young persons at the education centre for health and care professions in St. Gallen (BZGS) by conducting screening instruments. Furthermore, the investigators aim to identify risk and protective factors for the mental health of vocational trainees in health and care professions.

These results are both essential for further research and educational practice. Moreover, results may maximise the chances of creating in future meaningful intervention for young persons in this specific setting.

DETAILED DESCRIPTION:
Background:

Young person's undergoing training in the health or social services sector are confronted with issues such as dying, illness and severe personal tragedies while they are still in the process of their own development. This can have serious effects on their mental health. During this time, vocational school is a central part of young persons' lives. The YouCoMent project will initiate a sustainable promotion and maintenance of mental health and thus preventively counteract the development of mental health conditions.

In order to meet the special challenges of vocational schools in the health sector, this study pursues the following objectives:

To assess the current state of mental health of young persons at the educational centre.

To identify individual risk and protective factors for the mental health of young persons.

Methods:

This study is the first part of the YouCoMent project, which will be carried out at the education centre for health and care professions in St. Gallen (BZGS), Switzerland between 2023 and 2026.It has approx. 150 educators. The number of trainees in basic training is about 2800.

Every person will be asked through the BZGS internal E-Mail distribution lists to participate. Beforehand, between 20 and 24 January 2023. Data collection will be conducted on T1: 26 January 2023 and T2: 24 January 2025. Participation in the study is voluntary. The data collection is going to be carried out using a self-administered online questionnaire. Data collection will be conducted in anonymous form.

The quantitative data will be analysed using descriptive and, where appropriate, exploratory statistics, as well as analysed with statistical software (SPSS). The statistical analyses are carried out by researchers at the University of Applied Sciences of Eastern Switzerland in St. Gallen.

ELIGIBILITY:
Inclusion Criteria:

* All trainees at the centre

Exclusion Criteria:

* under age of 14

Ages: 14 Years to 64 Years | Sex: All
Age Groups: Child, Adult
Study Population: Sample of trainees in the health and social professions. Healthcare Assistant, Federal Diploma of Vocational Education and Training (FAGE), Certified Social Care Worker, Federal Diploma of Vocational Education and Training, Specialisation in people with disabilities (FABB), Certified Social Care Worker, Federal Diploma of Vocational Education and Training, Specialisation in children (FABK), Medical Practice Assistant (MPA), Dental assistant (DA), Health and Social Assistant (AGS), Registered Nurse (HF), Biomedical Analyst (BMA), Registered Operation Room Technician, Advanced Federal Diploma of Higher Education (OT).
  Sample of educators who teach in the aforementioned professions. No limitations are to be made regarding age, professional experience or duration of training.
Sampling Method: Non-Probability Sample
Enrollment: 2950 (Estimated)
Dates: Start 2023-01-26 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Patient Health Questionnaire at 2 years | T1: 20. January - 28. of February 2023 and T2: 24 January 2025 - 28. of February 2025
  Self-assessment instrument for the screening of the most common mental condition.
  Somatoform Disorder if >3 of 1a-m bother the patient "a lot". Major Depressive Syndrome if 2a or b and >5 of 2a-i are at least "More than half the days" Other Depressive Syndrome if 2a or b and >4 of 2a-i are at least "More than half the days" Panic Syndrome if 3a-d are "YES" and >4 of 4a-k are "YES" Other Anxiety Syndrome if 5a and >3 of 5b-g are "More than half the days" Bulimia Nervosa if 6a,b, and c and 8 are "YES" Binge Eating Disorder the same but 8 is either "NO" or left blank Alcohol abuse if any of 10a-e are "YES"
  Depression Severity. Total score for 9 items ranges from 0 to 27. Higher values indicate higher depressive symptom burden.
  Somatic Symptom Severity. Total score for 15 items ranges from 0 to 30. Higher values indicate higher somatic symptom burden.
  Stress. Total score for 10 items ranges from 0 - 20. Higher values indicate higher stress.

SECONDARY OUTCOMES:
Change from Baseline Self-Efficacy Scale at 2 years | T1: 20. January - 28. of February 2023 and T2: 24 January 2025 - 28. of February 2025
  The scales can be used to record convictions of subjective controllability or competence expectations in different demanding situations, namely for school and general life. The individual test score is obtained by adding up all ten items resulting in a score between 10 and 40. High values indicate a high general self-efficacy expectation.
Change from Baseline World Health Organization Disability Assessment Schedule 2.0 at 2 years | T1: 20. January - 28. of February 2023 and T2: 24 January 2025 - 28. of February 2025
  A generic assessment instrument for health and disability. The six domain scores are summed and converted into a summary score, which assumes a score between 0 and 100 (where 0 = no disability; 100 = full disability).
Change from Baseline Stress- and Coping-Inventory at 2 years | T1: 20. January - 28. of February 2023 and T2: 24 January 2025 - 28. of February 2025
  The Stress- and Coping-Inventory is a scientific questionnaire used to determine the current perceived stress and stress symptoms as well as to assess how people cope with stress with the help of coping strategies. It comprises 10 scales with 54 items The current perceived stress is measured with 3 scales consisting of 7 items each, ranging from 1 = not stressed to 7 = very stressed. With a range of 7 - 49, higher values indicate higher stress. The scale with the current total stress is the sum of the three stress scales. With a range of 21 - 147, higher values indicate higher stress.
  The physical and psychological stress symptoms are measured with 13 items from 1 = strongly disagree to 4 = strongly agree. With a range of 13 - 52, higher values indicate higher stress.
  Coping strategies are assessed with 5 scales of 4 items each, ranging from 1 = strongly disagree to 4 strongly agree. With a range of 4 - 16. Higher values indicate more effective stress coping.
Change from Baseline World Health Organization - assessment of self-rated health status at 2 years | T1: 20. January - 28. of February 2023 and T2: 24 January 2025 - 28. of February 2025
  One question assessing self-rated health status, formulated as "In general, how would you rate your health today," with the possible choices being "very good" (1), "good" (2), "moderate" (3), "bad" (4) or "very bad" (5)
Change from Baseline World Health Organization - current use of mental health services at 2 years | T1: 20. January - 28. of February 2023 and T2: 24 January 2025 - 28. of February 2025
  One question assessing current use of mental health services, formulated as "Have you been in treatment for a mental health condition in the last 12 months?" 1 = yes, 2 = no
Change from Baseline World Health Organization - perceived need for mental health services at 2 years | T1: 20. January - 28. of February 2023 and T2: 24 January 2025 - 28. of February 2025
  One question assessing perceived need for mental health services, formulated as "During the past 12 months, have you thought you might need help for psychological problems, your emotional problems, or alcohol or drug use?" 1 = yes, 2 = no
Change from Baseline Community-Attitude-toward-the-Mental-Ill (CAMI)-Inventory at 2 years | T1: 20. January - 28. of February 2023 and T2: 24 January 2025 - 28. of February 2025
  The Community Attitude to Mental Illness Inventory (CAMI) assess a respondent's attitude toward mental illness. With 40 Likert-scaled items (1 = Strongly agree - 5 = Strongly disagree) resulting in 4 dimensions (exclusion, integration, benevolence, social control). High scores on the subscales integration (10 items) and benevolence (10 items) reflect positive attitudes like support and tolerance, whereas high scores on the sub-dimensions exclusion (10 items) and social control (10 items) indicate stigmatizing attitudes.
Change from Baseline Sentiments, Attitudes and Concerns about Inclusive Education - Revised at 2 years | T1: 20. January - 28. of February 2023 and T2: 24 January 2025 - 28. of February 2025
  The instrument assesses views and concerns about inclusive education with the scales (1) Negative attitudes towards impairment, (2) Positive attitudes towards inclusive education, (3) Concerns about the concrete implementation of inclusive education consisting of each 5 items (1 = strongly disagree to 5 = strongly agree) With a range of 3 - 15. Higher values indicate more positive attitudes.
Change from Baseline Teacher Effectiveness in Inclusive Education at 2 years | T1: 20. January - 28. of February 2023 and T2: 24 January 2025 - 28. of February 2025
  The instrument assesses subjective effectiveness in inclusive education with the scales (1) Efficacy to use inclusive instructions (2) Efficacy in collaboration and (3) Efficacy in managing behaviour consisting of each 6 items (1 = strongly disagree to 6 = strongly agree). With a range of 3 - 18. Higher values indicate higher subjective efficacy for inclusive education.

CONTACTS AND LOCATIONS:
Overall Officials: Manuel P. Stadtmann, Prof. Dr., Principal Investigator — Competence Center for Mental Health - Eastern Switzerland
Locations (1):
- Competence Center for Mental Health, Sankt Gallen, Canton of St. Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Project homepage — https://www.youcoment.com/